CLINICAL TRIAL: NCT05621161
Title: Comparison of Ultrasound-Guided Lumbar Erector Spinae Plane Block And Fascia Iliaca Compartment Block for Pain Management Following Total Hip Prosthesis Surgery
Brief Title: ESPB vs FICB for Pain Management Following Total Hip Prosthesis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mursel Ekinci (Other Government)
Responsible Party: Sponsor-Investigator, Mursel Ekinci, Principal Investigator, Bursa City Hospital
Organization: Bursa City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BursaCityH1
Record Dates: First submitted 2022-11-07; First posted 2022-11-17 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis; Knee Disease; Knee Arthritis
Keywords: Total hip prosthesis surgery; Postoperative analgesia; Erector spina plan block; Fascia iliaca compartment block
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Fascia iliaca compartment block (FICB) group, and Erector spinae plane block (ESPB) group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupFICB= fascia iliaca compartment block (Active Comparator): ESP block will be performed. US probe will be placed longitudinally 2-3 cm lateral to the L3 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle (100 mm, 22G) will be inserted cranio-caudal direction and then for correction of the needle 2 ml saline will be injected deep into the erector spinae muscle fascia. Following confirmation of the correct position of the needle 30 ml 0.25% bupivacaine will be administered for the block.
  Interventions: Drug: Postoperative analgesia management
- Group ESPB = erector spina plan block (Active Comparator): FIC block will be performed in the supine position. The linear probe is placed transversely to identify the femoral artery, iliopsoas muscle, and fascia iliaca at the inguinal crease. The probe will be tilted cranially and caudally until optimal images of the fascia iliaca are obtained. Block needle (50 mm, 22G) will be passed through the iliac fascia via the in-plane method. Once the needle tip will be placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 2 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine 30 mL will be injected.
  Interventions: Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: Postoperative analgesia management — Intravenous paracetamol 1 gr and a dose of 0,5 mg/kg-1 tramadol intravenously will be performed on all patients 30 min before the end of the surgery for postoperative analgesia. Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. A patient-controlled device prepared with 5 mg/ ml tramadol will be attached to all patients with a protocol including 10 mg bolus without infusion dose, 10 min lockout time, and 4-hour limit. If the VAS score will be ≥ 4, 0,5 mg/kg-1 meperidine IV will be administered.

SUMMARY:
Hip arthroplasty surgery is frequently performed on elderly patients in the community and it is associated with long-term postoperative hospital stays and high mortality.

Postoperative pain management is a multimodal process that includes intravenous and regional anesthesia methods. The ultrasound(US) guided erector spinae plane block (ESPB) is injected with a local anesthetic into the deep fascia of the erector spinae. In the literature, it has been reported that ESPB provides effective analgesia after a hip surgery. The fascia iliaca compartment block (FICB) is a safe method used for postoperative analgesia following hip, femoral, and knee surgeries.

The aim of this study is to compare US-guided FICB and ESPB for postoperative analgesia management after total hip prosthesis surgery.

DETAILED DESCRIPTION:
Hip arthroplasty surgery is frequently performed on elderly patients in the community and it is associated with long-term postoperative hospital stays and high mortality. Severe postoperative pain may further reduce the limited cardiopulmonary capacity, especially in the elderly population. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Postoperative pain management is a multimodal process that includes intravenous and regional anesthesia methods. Parenteral opioids are generally preferred in the management of acute postoperative pain. However, opioids have undesired adverse events such as nausea, vomiting, itching, sedation, and respiratory depression (opioid-related adverse events). Regional anesthesia techniques are frequently preferred as a part of multimodal analgesia in hip surgeries. Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment. US-guided interfascial plane blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice.

The ultrasound(US) guided erector spinae plane block (ESPB) is injected with a local anesthetic into the deep fascia of the erector spinae. Visualization of sonoanatomy with the US is simple and the spread of local anesthetic solution can be seen easily in the deep fascia of the erector spinae. Visualization of sonoanatomy in the US is easy, and the spread of local anesthetic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves. In the literature, it has been reported that ESPB provides effective analgesia after a hip surgery. The fascia iliaca compartment block (FICB) is a safe method used for postoperative analgesia following hip, femoral, and knee surgeries.

The aim of this study is to compare US-guided FICB and ESPB for postoperative analgesia management after total hip prosthesis surgery. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), and adverse effects related to opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III
* Aged 18-80 years
* Who will be scheduled for total hip prosthesis surgery under spinal anesthesia

Exclusion Criteria:

* Patients who have a history of bleeding diathesis
* Take anticoagulant therapy
* History of chronic pain before surgery
* Known local anesthetics and opioid allergy
* Pregnancy or lactation
* Infection at the site of block
* Patients who do not accept the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The tramadol consumption on PCA device will be evaluated

SECONDARY OUTCOMES:
Postoperative pain score | Postoperative 1, 2, 4, 8, 16 and 24 hours
  Postoperative pain assessment will be performed using the Numerical Rating Scale (0 = no pain, 10 = the most severe pain felt)

CONTACTS AND LOCATIONS:
Locations (1):
- Mursel Ekinci, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Gao Y, Tan H, Sun R, Zhu J. Fascia iliaca compartment block reduces pain and opioid consumption after total hip arthroplasty: A systematic review and meta-analysis. Int J Surg. 2019 May;65:70-79. doi: 10.1016/j.ijsu.2019.03.014. Epub 2019 Mar 25. PMID 30922995
- [Background] Tulgar S, Senturk O. Ultrasound guided Erector Spinae Plane block at L-4 transverse process level provides effective postoperative analgesia for total hip arthroplasty. J Clin Anesth. 2018 Feb;44:68. doi: 10.1016/j.jclinane.2017.11.006. Epub 2017 Nov 14. No abstract available. PMID 29149734
- [Background] Deniz S, Atim A, Kurklu M, Cayci T, Kurt E. Comparison of the postoperative analgesic efficacy of an ultrasound-guided fascia iliaca compartment block versus 3 in 1 block in hip prosthesis surgery. Agri. 2014;26(4):151-7. doi: 10.5505/agri.2014.76993. PMID 25551810
- [Derived] Kaciroglu A, Ekinci M, Dikici M, Aydemir O, Demiroluk O, Erdogan D, Golboyu BE, Alver S, Ciftci B, Gurbuz H. Lumbar erector spinae plane block versus infrainguinal fascia iliaca compartment block for pain management after total hip arthroplasty: a randomized clinical trial. Pain Med. 2024 Apr 3;25(4):257-262. doi: 10.1093/pm/pnad166. PMID 38127974